CLINICAL TRIAL: NCT05001698
Title: A Phase I, Open-label, Single-Arm, Multiple-Dose Study to Evaluate the Pharmacokinetics, Safety and Tolerability of Anifrolumab in Chinese Participants With Systemic Lupus Erythematosus (SLE)
Brief Title: Anifrolumab PK Study for Systemic Lupus Erythematosus (SLE)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D3468C00002
Record Dates: First submitted 2021-06-30; First posted 2021-08-12 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Systemic Lupus Erythematosus
Keywords: systemic lupus erythematosus; SLE; pharmacokinetic; anifrolumab
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — anifrolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anifrolumab (Experimental): All eligible participants will receive anifrolumab via intravenous (IV) infusion pump.
  Interventions: Biological: Anifrolumab

INTERVENTIONS:
Biological: Anifrolumab — intravenous infusion (IV)

SUMMARY:
To assess the pharmacokinetic parameters of anifrolumab in Chinese participants with active systemic lupus erythematosus(SLE).

DETAILED DESCRIPTION:
This is a Phase I, open-label, single-arm, multiple-dose study to evaluate the pharmacokinetics (PK), pharmacodynamics(PD), safety and tolerability profile of intravenously administered anifrolumab in Chinese participants with active SLE despite receiving standard of care (SOC).

ELIGIBILITY:
Key inclusion criteria:

1. Aged 18 to 60 years.
2. Body weight ≥ 40 kg.
3. Confirmed diagnosis of SLE(1997 ACR revised criteria) for ≥ 24 weeks.
4. Must be receiving at least one of the following SOC regimens at screening:

   1. oral prednisone monotherapy: ≥ 7.5 mg/day and ≤ 40 mg/day, stable for > 2 weeks;
   2. Immunosuppressant(s) with or without OCS: antimalarials, AZA, MMF, MTX, mizoribine permitted; stable for ≥ 8 weeks; maximum dose required;
   3. Oral prednisone plus immunosuppressant: start date, stability and maximum dose required.
5. At least one of these antibodies positive: ANA, anti-dsDNA and anti-Smith.
6. At screening, SLEDAI-2K score ≥ 6 points.
7. Chest imaging shows no clinically significant abnormalities (unless due to SLE).
8. No evidence or medical history of active TB, indeterminate TB should be referred to a TB specialist.
9. All participants should use effective contraception methods as protocol requests.

Key exclusion criteria:

1. History or current diagnose of clinically significant non-SLE related vasculitis, severe or unstable neuropsychiatric SLE, active severe SLE-driven renal disease, catastrophic anti-phospholipid syndrome, inflammatory joint or skin disease other than SLE, non-SLE disease that has required treatment of certain dosage of corticosteroid.
2. History or evidence of suicidal ideation or suicidal behavior.
3. History or current diagnose of MTCD or overlap syndrome, unless overlap with RA or MTCD which has developed into SLE.
4. History of recurrent infection requiring hospitalization and IV antibiotics, or opportunistic infection requiring hospitalization or IV antimicrobial treatment within 3 years of randomization, or clinically significant chronic infection within 3 months, or recent infection still under treatment.
5. History of immunodeficient condition, HIV positive included.
6. Confirmed HBsAg positive, or HBcAb positive and HBV DNA detectable.
7. History of severe case of herpes zoster.
8. Herpes zoster, CMV or EB infection which has not completely resolved within 12 weeks before screening.
9. Acute COVID-19 infection or history of severe COVID-19.
10. History of cancer, apart from cured squamous or basal cell carcinoma and cervical cancer in situ.
11. Women participants with abnormal pap smear results.
12. Prior receipt of anifrolumab ,or any commercially available biologic agent, or protein kinase inhibitor or any investigational product within 5 half-lives, including B cell-depleting therapy, belimumab, JAK or BTK inhibitor.
13. Known history of allergy to any component of the IP formulation or protein related products.
14. Receipt of any of the following:

    1. Intramuscular or IV glucocorticosteroids within 6 weeks;
    2. Any live or attenuated vaccine within 8 weeks;
    3. Any restricted medication listed in protocol;
    4. Blood transfusion within 4 weeks.
15. Certain laboratory test results requirements.
16. Concurrent enrolment in another clinical study.
17. History or current alcohol, drug or chemical abuse within 1 year.
18. Major surgery within 8 weeks or planned elective major surgery.
19. Blood donation or blood loss more than 400 mL within 3 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-06-02 (Actual)

PRIMARY OUTCOMES:
Time to maximum observed plasma concentration (Tmax) of anifrolumab. | Day 1 to Day 141
  To characterise the pharmacokinetic (PK) profile of anifrolumab via intravenous (IV) infusion.
Maximum observed plasma concentration (Cmax) of anifrolumab. | Day 1 to Day 141
  To characterise the pharmacokinetic (PK) profile of anifrolumab via intravenous (IV) infusion.
Area under plasma concentration-time curve over dosing interval (AUC[tau]) of anifrolumab. | Day 1 to Day 141
  To characterise the pharmacokinetic (PK) profile of anifrolumab via intravenous (IV) infusion.
Pre-dose trough concentration (Ctrough) of anifrolumab. | Day 1 to Day 141
  To characterise the pharmacokinetic (PK) profile of anifrolumab via intravenous (IV) infusion.
The volume of plasma cleared of drug per unit time (CL) of anifrolumab. | Day 1 to Day 141
  To characterise the pharmacokinetic (PK) profile of anifrolumab via intravenous (IV) infusion.

SECONDARY OUTCOMES:
Incidence of adverse events | From Screening, Day 1 to Day 141
  To characterise the safety and tolerability of anifrolumab via IV infusion.
Incidence of abnormal vital signs | From Screening, Day 1 to Day 141
  To characterise the safety and tolerability of anifrolumab via IV infusion.
Incidence of abnormal laboratory parameters | Day 29, 57, 85, 113, 141
  To characterise the safety and tolerability of anifrolumab via IV infusion.
Anti-drug antibodies (ADA) | Day 1, 85, 113, 141
  To characterise the immunogenicity of anifrolumab via IV infusion.
21-gene Type I interferon PD signature | Screening, Day 29, 85, 113, 141
  To evaluate the IFN level change from baseline after administration of anifrolumab.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Research Site, Nantong
  - Research Site, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home